CLINICAL TRIAL: NCT00555828
Title: A Phase 1b/2a Dose Escalation Study to Assess the Safety and Feasibility of Transendocardial Delivery of 3 Different Doses of Allogeneic Mesenchymal Precursor Cells (MPCs) in Subjects With Recent Acute Myocardial Infarction
Brief Title: Safety Study of Allogeneic Mesenchymal Precursor Cells (MPCs) in Subjects With Recent Acute Myocardial Infarction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Angioblast Systems (Industry)
Responsible Party: Donna Skerrett, MD ; Medical Director, Angioblast Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMT-AB001
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2009-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Myocardial infarct; Infarction
MeSH Terms: conditions — Myocardial Infarction; Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A1 (Experimental): 5 subjects randomized to receive 25 M allogeneic MPCs by transendocardial injection
  Interventions: Genetic: Allogeneic Mesenchymal Precursor Cells (MPCs)
- A2 (Other): 5 subjects randomized to receive standard-of-care treatment with NOGA® mapping and staged injections.
  Interventions: Procedure: Standard-of-care treatment with NOGA® mapping and staged injections.
- B1 (Experimental): 5 subjects randomized to receive 75 M allogeneic MPCs by transendocardial injection
  Interventions: Genetic: Allogeneic Mesenchymal Precursor Cells (MPCs)
- B2 (Other): 3 subjects randomized to receive standard-of-care treatment with NOGA® mapping and staged injections.
  Interventions: Procedure: Standard-of-care treatment with NOGA® mapping and staged injections.
- C1 (Experimental): 5 subjects randomized to receive 150 M allogeneic MPCs by transendocardial injection
  Interventions: Genetic: Allogeneic Mesenchymal Precursor Cells (MPCs)
- C2 (Other): 2 subjects randomized to receive standard-of-care treatment with NOGA® mapping and staged injections.
  Interventions: Procedure: Standard-of-care treatment with NOGA® mapping and staged injections.

INTERVENTIONS:
Genetic: Allogeneic Mesenchymal Precursor Cells (MPCs) — 25 M allogeneic MPCs by transendocardial injection
  Arms: A1
Procedure: Standard-of-care treatment with NOGA® mapping and staged injections. — Standard-of-care treatment with NOGA® mapping and staged injections.
  Arms: A2
Genetic: Allogeneic Mesenchymal Precursor Cells (MPCs) — 75 M allogeneic MPCs by transendocardial injection
  Arms: B1
Procedure: Standard-of-care treatment with NOGA® mapping and staged injections. — Standard-of-care treatment with NOGA® mapping and staged injections.
  Arms: B2
Genetic: Allogeneic Mesenchymal Precursor Cells (MPCs) — 150 M allogeneic MPCs by transendocardial injection
  Arms: C1
Procedure: Standard-of-care treatment with NOGA® mapping and staged injections. — Standard-of-care treatment with NOGA® mapping and staged injections.
  Arms: C2

SUMMARY:
Primary Objective The primary objective of this study is to evaluate the safety and feasibility of transendocardial injection using the Cordis Biosense NogaStarTM Mapping Catheter with the Biosense MyostarTM Left Ventricular Injection Catheter of 25 M, 75 M, and 150 M allogeneic mesenchymal precursor cells (MPCs) in subjects with AMI.

SecondaryObjective

The secondary objectives are to explore functional efficacy for subsequent study design, as well as late-term dose related tolerance, by:

* Evaluating the effect of allogeneic MPCs on exploratory efficacy endpoints related to cardiac function on Days 90, 180, and 1 year
* Evaluating the change from baseline in the Medical Outcome Study Short Form (SF-36), Kansas City Cardiomyopathy Questionnaire, Seattle Angina Questionnaire, and the New York Heart Association Classification at 30 days, 3 and 6 months, and 1, 2, and 3 years
* Evaluating follow-up safety through Day 360
* Providing preliminary data to support dose selection for future studies

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. An ST-elevation MI (STEMI) within 2 to 10 days of study enrollment. The STEMI must be documented by ECG with ST-segment elevation >1 mm in at least 2 contiguous precordial leads or in at least 2 adjacent limb leads. If there is a history of a previous AMI prior to the qualifying MI, then there must be a documented EF ≥ 50% by 2D echocardiogram within 12 months of enrollment.
3. Successful percutaneous revascularization with Thrombolysis in Myocardial Infarction (TIMI)-3 flow of the infarct-related artery.
4. A baseline 2D echocardiogram with EF ≥ 30 and ≤ 50% following PCI.
5. Creatinine level ≤ 1.5mg/dL within 24 hours of study procedure.
6. Hematocrit ≥ 30% within 24 hours of study procedure.
7. White Blood Cell count < 20k/mm3 within 24 hours of study procedure.
8. Platelet count ≥ 100k/mm3 within 24 hours of study procedure.
9. INR ≤ 1.7 within 24 hours of study procedure.
10. Total bilirubin <3 mg/dL, albumin >2.8 g/dL, aspartate aminotransferase(AST) ≤ 2.5x the upper limit of normal, gamma glutamyltranspeptidase (GGT) ≤ 1.5 x the upper limit of normal.
11. If the subject or partner is of childbearing potential, he or she must be willing to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening and for a period of at least 16 weeks after surgery.
12. Female subjects of childbearing potential must have a negative serum pregnancy test at screening (within 2 weeks of enrollment) and a negative serum or urine pregnancy test on the day of cell implantation.
13. Willing and able to understand, sign, and date the Informed Consent Form (ICF).
14. Must be willing to return for required follow-up visits.
15. Must be able to follow postoperative management program.

Exclusion Criteria:

1. Subject is hemodynamically unstable at Day 5 post-AMI as demonstrated by any of the following:

   1. Killip Class 4 indicative of cardiogenic shock.
   2. Requirement of intra-aortic balloon pump or IV inotropic support for the maintenance of mean arterial blood pressure ≥ 60 mmHg.
2. Sustained ventricular tachycardia as demonstrated by QRS complexes wider than 120 msec, lasting >30 secs, and >100 bpm occurring >48 hours following PCI without any identifiable, reversible cause (ie, electrolyte imbalance).
3. Further revascularization planned for the next 30 days.
4. Chronic atrial fibrillation.
5. A wall thickness in the target region <8 mm as determined by 2D echocardiography(the target region is defined at the time of NOGA® mapping).
6. An LV thrombus.
7. Severe peripheral vascular disease precluding femoral artery access as determined at time of original catheterization.
8. Aortic stenosis as determined as valve area less than 1 cm2 that prohibits catheter access to the LV.
9. Echocardiographic evidence of hypertrophic cardiomyopathy indicating heart muscle thickness >15 mm.
10. Human immunodeficiency virus (HIV)
11. Serum glucose level ≥ 400 mg/dl within 24 hours of study procedure
12. Serum glucose level 300-400 mg/dl and presence of urine ketones within 24 hours of study procedure.
13. Claustrophobic, or with medical conditions or contradictions that impede performing baseline MRI study.
14. An active uncontrolled infection.
15. A prosthetic aortic valve.
16. Presence of ≥ 20% anti-HLA antibody titers and/or having antibody specificities to donor HLA antigens.
17. A current or prior history within the last 3 years of neoplasm (excluding basal cell) and/or any active neoplasm within the last 24 months.
18. A known hypersensitivity to dimethyl sulfoxide (DMSO), murine and/or bovine products.
19. Pregnancy or breastfeeding.
20. Imprisoned at the time of enrollment.
21. A treatment and/or an uncompleted follow-up treatment of any investigational therapy within 6 months before implantation surgery and intent to participate in any other investigational drug or cell therapy study during the 3-year follow-up period of this study.
22. Active participation in other research therapy for cardiovascular repair/regeneration.
23. A prior recipient of stem precursor cell therapy for cardiac repair.
24. Any medical condition that would affect the investigator's ability to evaluate the subject's condition or could compromise the subject's safety.
25. Any condition that, in the judgment of the investigator, would prohibit the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and feasibility of transendocardial injection using the Cordis Biosense NogaStarTM Mapping Catheter with the Biosense MyostarTM Left Ventricular Injection Catheter of allogeneic mesenchymal precursor cells (MPCs) in subjects with AMI. | 30 days

SECONDARY OUTCOMES:
Explore efficacy for subsequent study design and dose related tolerance: •Effect related to cardiac function.•Change from baseline in SF-36, KCCQ, SAQ, and the NYHA Classification.•Follow-up safety through Day 360 • Dose selection for future stu | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emerson C. Perin, MD, PhD, Principal Investigator — Texas Heart Institute/St. Luke's Hospital
Locations (2):
- United States (2):
  - University of Minnesota/Minneapolis Heart Institute, Minneapolis, Minnesota
  - Texas Heart Institute/St. Luke's Hospital, Houston, Texas